CLINICAL TRIAL: NCT05551039
Title: RegoFlex EU/Real World Evidence on Stivarga Flexible Dosing in Patients With Metastatic Colorectal Cancer in Europe
Brief Title: An Observational Study, Called RegoFlex EU, to Learn More About the Use of Stivarga at Reduced Doses as Recommended (Flexible Dosing) to Treat People With Metastatic Colorectal Cancer in Real World Settings in Europe
Acronym: RegoFlex EU
Status: Completed | Type: Observational
Sponsor: Bayer (Industry)
Responsible Party: Sponsor
Other Study IDs: 22124
Record Dates: First submitted 2022-08-26; First posted 2022-09-22 (Actual); Last update posted 2023-01-26 (Actual); Status verified 2023-01

CONDITIONS: Metastatic Colorectal Cancer
MeSH Terms: conditions — Colorectal Neoplasms

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Physicians treating patients with mCRC: Physicians provide case histories of mCRC patients
  Interventions: Other: Retrospective patient chart review

INTERVENTIONS:
Other: Retrospective patient chart review — Retrospective patient chart review to be completed by mCRC-treating physicians. Data is collected through an online case report form (CRF); physicians provide case histories of mCRC patients who initiated regorafenib treatment in most recent 3 years (2019-2021).

SUMMARY:
This is an observational study in which data from patients with metastatic colorectal cancer in three European countries who received STIVARGA® (regorafenib), are collected. In observational studies, only observations are made without specified advice or interventions.

Metastatic colorectal cancer (mCRC) is a cancer that starts in the large bowel or the rectum (the lowest part of the gut) and has spread to other parts of the body. Regorafenib is an anti-cancer drug that blocks several proteins called enzymes, which are involved in the development and growth of cancer. A wide range of such enzymes called tyrosine kinases are targeted.

In 2013, regorafenib was approved in Europe for doctors to prescribe to people with mCRC who have previously been treated or cannot receive other available treatments. It is known that doctors may change/reduce the amount (the dose) of regorafenib they give (flexible dosing), so that the patients better tolerate the treatment. However, little information is available on the doses of regorafenib given in France, Italy, and Belgium in usual practice.

In this study researchers want to learn more about how and in which amount regorafenib is usually given to patients with mCRC in France, Italy, and Belgium:

* at the beginning
* during, and
* at the end of the regorafenib therapy.

In addition, the study team will collect data about/if:

* the treatment duration at each treatment dose of regorafenib,
* the number of people who received reduced initial dosing of regorafenib in real word settings in France, Italy, and Belgium,
* reduced (flexible) initial dosing of regorafenib allows patients to stay longer on treatment.

To answer these questions, the researchers will look back at cases that have already happened when the study begins. The data will be collected through an online case report form. The doctors will provide case histories of mCRC patients who started regorafenib treatment in most recent 3 years and 4 months (from January 1, 2019 to Apr 30, 2022) or up until 3 months prior to the date of data collection.

Besides this data collection, no further tests or examinations are planned in this study.

There are no required visits or tests in this study.

ELIGIBILITY:
Inclusion Criteria:

* Patients with a histopathological or cytological diagnosis of colorectal cancer and metastatic disease (stages IVA, IVB, or IVC)
* Patients must have initiated regorafenib as monotherapy, regardless of line of therapy, from January 1, 2019 to December 31, 2021 (or up until 3 months prior to date of data collection, whichever occurs latest)
* Aged ≥18 years at index date

Exclusion Criteria:

* Patients with regorafenib treatment prior to January 1, 2019
* Patients who have participated in a clinical trial

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients with mCRC in France, Italy and Belgium and initiated regorafenib therapy between January 1, 2019 and December 31, 2021
Sampling Method: Non-Probability Sample
Enrollment: 300 (Actual)
Dates: Start 2022-08-15 (Actual); Primary Completion 2023-01-15 (Actual); Study Completion 2023-01-15 (Actual)

PRIMARY OUTCOMES:
Proportion of patients initiating a flexible regorafenib dose (40, 80, or 120 mg) versus 160 mg | Retrospective analysis from 01-Jan-2019 up to 30-Apr-2022 (or up until 3 months prior to date of data collection, whichever occurs latest)
Dose at treatment end (last prescribed regorafenib dose): 40, 80, 120, or 160 mg | Retrospective analysis from 01-Jan-2019 up to 30-Apr-2022 (or up until 3 months prior to date of data collection, whichever occurs latest)
Average dose intensity at first and subsequent cycles | Retrospective analysis from 01-Jan-2019 up to 30-Apr-2022 (or up until 3 months prior to date of data collection, whichever occurs latest)
  The sum of dose strength (mg) will be divided by the days on therapy in each cycle.
Time to first dose change | Retrospective analysis from 01-Jan-2019 up to 30-Apr-2022 (or up until 3 months prior to date of data collection, whichever occurs latest)
  Time to first dose change: time (months) from date of initial regorafenib dose to 1st dose increase/decrease among patients initiating a flexible regorafenib dose (40, 80, or 120 mg)
Time to first full dose of 160 mg | Retrospective analysis from 01-Jan-2019 up to 30-Apr-2022 (or up until 3 months prior to date of data collection, whichever occurs latest)
  Time to 1st full dose of 160 mg: time (months) from date of initial regorafenib dose to 1st full dose of 160 mg during the treatment history among patients with 40, 80, or 120 mg initial dose, overall and by initial dose.
Number of cycles received | Retrospective analysis from 01-Jan-2019 up to 30-Apr-2022 (or up until 3 months prior to date of data collection, whichever occurs latest)
Proportion of patients initiating 1, 2, 3, or more cycles | Retrospective analysis from 01-Jan-2019 up to 30-Apr-2022 (or up until 3 months prior to date of data collection, whichever occurs latest)
  The label recommended regorafenib treatment cycle is 28 days.
Duration of treatment (DoT) | Retrospective analysis from 01-Jan-2019 up to 30-Apr-2022 (or up until 3 months prior to date of data collection, whichever occurs latest)
  Duration of treatment: time (months) from date of initial regorafenib dose to date of last dose prior to a >2-week gap during the follow up period.
Time to discontinuation (TTD) | Retrospective analysis from 01-Jan-2019 up to 30-Apr-2022 (or up until 3 months prior to date of data collection, whichever occurs latest)
  Time to discontinuation: time (months) from date of initial regorafenib dose to date of discontinuation (as indicated by CRF)
Proportion of patients with reasons for discontinuation | Retrospective analysis from 01-Jan-2019 up to 30-Apr-2022 (or up until 3 months prior to date of data collection, whichever occurs latest)
  Reasons for discontinuation includes: distant progression/relapse, local progression/relapse, patient choice to discontinue therapy, poor performance status, side effects, new primary malignancy, death, lost to follow up, coronavirus disease 2019 (COVID-19)-related and other.

SECONDARY OUTCOMES:
Descriptive summary of demographics characteristics | Retrospective analysis from 01-Jan-2019 up to 30-Apr-2022 (or up until 3 months prior to date of data collection, whichever occurs latest)
  Demographic characteristics includes: age, sex, index year (calendar year of regorafenib treatment initiation date), race, alive or deceased at time of data collection, primary cause of death (for deceased patients only).
Descriptive summary of Stage of disease | Retrospective analysis from 01-Jan-2019 up to 30-Apr-2022 (or up until 3 months prior to date of data collection, whichever occurs latest)
  Stage of disease includes: Stage IVA; Stage IVB and Stage IVC
Descriptive summary of Eastern Cooperative Oncology Group (ECOG) performance status | Retrospective analysis from 01-Jan-2019 up to 30-Apr-2022 (or up until 3 months prior to date of data collection, whichever occurs latest)
  ECOG scale scores are: 0, 1, 2, 3, 4 and Unknow. The higher score means worse performance status.
Descriptive summary of Primary tumor status | Retrospective analysis from 01-Jan-2019 up to 30-Apr-2022 (or up until 3 months prior to date of data collection, whichever occurs latest)
  Primary tumor status includes: Local recurrence; Resected and Unresected
Descriptive summary of Number of metastatic | Retrospective analysis from 01-Jan-2019 up to 30-Apr-2022 (or up until 3 months prior to date of data collection, whichever occurs latest)
  Number of metastatic includes: 1, 2 and ≥3
Descriptive summary of Site of metastasis | Retrospective analysis from 01-Jan-2019 up to 30-Apr-2022 (or up until 3 months prior to date of data collection, whichever occurs latest)
  Site of metastasis includes: Bone, Liver, Lung, Lymph node, Peritoneum and Other.
Descriptive summary of K-RAS mutation status and N-RAS mutation status | Retrospective analysis from 01-Jan-2019 up to 30-Apr-2022 (or up until 3 months prior to date of data collection, whichever occurs latest)
  K-RAS mutation status and N-RAS mutation status includes: Wild type, Mutated and Unknown.
Descriptive summary of Line of therapy (LOT) for regorafenib | Retrospective analysis from 01-Jan-2019 up to 30-Apr-2022 (or up until 3 months prior to date of data collection, whichever occurs latest)
  Line of therapy (LOT) for regorafenib includes: 2nd, 3rd, 4th and 5th or higher.
Descriptive summary of Prior adjuvant treatment | Retrospective analysis from 01-Jan-2019 up to 30-Apr-2022 (or up until 3 months prior to date of data collection, whichever occurs latest)
  Prior adjuvant treatment includes: No and Yes.
Descriptive summary of Treatments prior to index date, overall and by LOT | Retrospective analysis from 01-Jan-2019 up to 30-Apr-2022 (or up until 3 months prior to date of data collection, whichever occurs latest)
  Treatments includes: Fluorouracil, Capecitabine, Irinotecan, Leucovorin, Mitomycin, Oxaliplatin, Anti-EGFR monoclonal antibody snf Anti-VEGF monoclonal antibody.
Descriptive summary of Pre-existing comorbidities | Retrospective analysis from 01-Jan-2019 up to 30-Apr-2022 (or up until 3 months prior to date of data collection, whichever occurs latest)
  Pre-existing comorbidities: Asthma, Atrial fibrillation, Auto-immune disease, Cardiac dysfunction, Chronic obstructive pulmonary disease, COVID-19, Diabetes, Hepatitis C, AIDS/HIV, Human papillomavirus, Liver dysfunction, Parkinson's, Peripheral neuropathy, Renal dysfunction, Thrombocytopenia, Venous thromboembolism, Other and None.

CONTACTS AND LOCATIONS:
Locations (1):
- Many locations, Whippany, New Jersey, United States

IPD SHARING:
Plan to Share IPD: No
Availability of this study's data will later be determined according to Bayer's commitment to the EFPIA/PhRMA "Principles for responsible clinical trial data sharing". This pertains to scope, timepoint and process of data access.
  As such, Bayer commits to sharing upon request from qualified researchers patient-level clinical trial data, study-level clinical trial data, and protocols from clinical trials in patients for medicines and indications approved in the US and EU as necessary for conducting legitimate research. This applies to data on new medicines and indications that have been approved by the EU and US regulatory agencies on or after January 01, 2014.
  Interested researchers can use www.clinicalstudydatarequest.com to request access to anonymized patient-level data and supporting documents from clinical studies to conduct research. Information on the Bayer criteria for listing studies and other relevant information is provided in the Study sponsors section of the portal.